CLINICAL TRIAL: NCT01252394
Title: ScO2 and Cardiac Output - Correspondence Study in Hemodialysis Patients
Brief Title: Correspondence of ScO2 and Cardiac Output in Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danish State Hospital (Other)
Responsible Party: Joakim Cordtz/MD, Department of Nephrology, Copenhagen University Hospital
Other Study IDs: ScO2 cardiac output
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-10

CONDITIONS: Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis patients

SUMMARY:
The study aims to investigate the correspondence between changes in central venous oxygen saturation (ScO2) and in cardiac output during hemodialysis. In 12 hemodialysis patients with an A-V fistula, a thoracic bioimpedance cardiograph will be validated for cardiac output measurements during ongoing hemodialysis. Provided this validation is satisfactory, impedance cardiography cardiac output and ScO2 will be measured at intervals during hemodialysis in 25 hemodialysis patients with a central vascular access. Absolute values and trends will be compared.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory hemodialysis patients in the Copenhagen University Hospital department of Nephrology.

Exclusion Criteria:

Age below 18 years. Failure to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Soeren D Ladefoged, MD, Study Director — Dep. of Nephrology, Copenhagen University Hospital.
Locations (1):
- Copenhagen University Hospital, Copenhagen E, Denmark

REFERENCES:
- [Background] Cordtz J, Olde B, Solem K, Ladefoged SD. Central venous oxygen saturation and thoracic admittance during dialysis: new approaches to hemodynamic monitoring. Hemodial Int. 2008 Jul;12(3):369-77. doi: 10.1111/j.1542-4758.2008.00283.x. PMID 18638095